CLINICAL TRIAL: NCT05602142
Title: A Phase 1/2 Study of [11C]CPPC as a Clinical PET Radioligand Biomarker of Microglial Activation in ALS
Brief Title: Study of [11C]CPPC as a Clinical PET Radioligand Biomarker of Microglial Activation in ALS
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00343494; W81XWH-22-1-0130 (Other Grant/Funding Number: Department Of Defense)
Record Dates: First submitted 2022-10-21; First posted 2022-11-01 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: ALS
Keywords: Biomarkers

STUDY DESIGN:
Intervention Model Description: Disease group and healthy controls will receive the same drug
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [11C]CPPC (Experimental): All participants will receive [11C]CPPC which is a radiotracer ligand that specifically binds to CSF1R.
  Interventions: Drug: [11C]CPPC PET ligand

INTERVENTIONS:
Drug: [11C]CPPC PET ligand — Radioactive PET ligand to determine microglia expression of colony stimulating factor 1 receptor (CSF1R).
  Other Names: 5-cyano-N-(4-(4-[11C]methylpiperazin-1-yl)-2-(piperidin-1-yl)phenyl)furan-2-carboxamide

SUMMARY:
1. Establish the safety and tolerability of the 5-cyano-N-(4-(4-[11C]Methylpiperazin-1-yl)-2-(Piperidin-1-yl)Phenyl)Furan-2-carboxamide ([11C]CPPC) PET radioligand in ALS patients and controls
2. Examine whether [11C]CPPC PET uptake is elevated in brains of ALS patients and whether there is a correlation with clinical phenotype.
3. Correlate [11C]CPPC PET imaging with other ALS outcome measures and biofluid biomarkers
4. Examine longitudinal changes in [11C]CPPC PET imaging during disease course.

DETAILED DESCRIPTION:
There are a paucity of reliable serum and cerebrospinal (CSF) biomarkers and validated neuroimaging techniques to aid in amyotrophic lateral sclerosis (ALS) diagnosis, prognosis, or pharmacodynamic insight. Positron emission tomography (PET) imaging is a technique that uses radioactive molecules attached to a ligand of interest which localizes to the desired target, allowing for visualization of the three dimensional distribution of the ligand's target receptor.

One of the upstream processes that are thought to lead to motor neuron degeneration in ALS is microglial dysfunction, resulting in the initiation of neuroinflammatory cascades. Macrophage colony stimulating factor 1 receptor (CSF1R) is found on microglia predominately in the brain, with low levels of expression in neurons and other neural cells, making it a promising target for studying microglial activation.

Given CSF1's potential role in ALS disease progression, and that its receptor (CSF1R) can be directly targeted, ligands binding this receptor are an area of interest for imaging in ALS. [11C]CPPC [5-cyano-N-(4-(4-[11C]methylpiperazin-1-yl)-2-(piperidin-1-yl)phenyl)furan-2-carboxamide], is a positron-emitting, high-affinity ligand that is specific for CSF1R.

The aims of this study are as follows:

1. Establish the safety and tolerability of the [11C]CPPC PET radioligand in ALS patients and controls
2. Examine whether [11C]CPPC PET uptake is elevated in brains of ALS patients and whether there is a correlation with clinical phenotype.
3. Correlate [11C]CPPC PET imaging with other ALS outcome measures and biofluid biomarkers
4. Examine longitudinal changes in [11C]CPPC PET imaging during disease course.

ELIGIBILITY:
Inclusion Criteria

1. Have the ability to understand the requirements of the study, provide written informed consent, understand and provide written authorization for the use and disclosure of Protected Health Information (PHI) [per Health Insurance Portability and Accountability Act (HIPAA) Privacy Ruling] and comply with the study procedures.
2. Men and women at least 18 years old.
3. Male patients, who have not had a vasectomy and a confirmed zero sperm count, must agree for the duration of the study to:

   * use a condom during sexual intercourse with female partners who are of reproductive potential AND to have female partners use an additional effective means of contraception (e.g., diaphragm plus spermicide, or oral contraceptives) OR
   * male patient must agree to abstain from sexual intercourse during the study
4. Women must have a negative serum pregnancy test and practice an acceptable method of contraception or be of non-childbearing potential (post-menopausal for at least 2 years or who have undergone hysterectomy, oophorectomy or surgical sterilization). Women must not be breastfeeding.
5. Geographic accessibility to the study center and the ability to travel to the clinic for study visits.
6. Presence of a willing and able caregiver.
7. Diagnosis of ALS based on examination by the site PI, meeting El Escorial criteria for possible, laboratory-supported probable, probable or definite ALS or be a person without a diagnosis of ALS disorder.
8. Vital capacity ≥ 50% of predicted normal for age, height and gender measured in the seated position and the ability to lie supine for a period of 1 hour.
9. Agrees to the visit schedule as outlined in the informed consent.
10. Pre-study labs within normal range, or if abnormal, deemed not clinically significant by the site investigator.

Exclusion Criteria:

1. Weakness due to causes other than ALS.
2. Receipt of any investigational drug, device or biologic within 10 days of administration of study compound.
3. Use of anti-inflammatory medications, immunosuppressants, or benzodiazepines within 7 days of administration of study compound.
4. Any concomitant medical disease or condition limiting the safety to participate including, but not limited to:

   1. Coagulopathy
   2. Active infection
5. Any condition that the site PI feels may interfere with participation in the study.
6. Inability to provide informed consent as determined by the site PI.
7. Known clinical evidence of frontotemporal dementia.
8. Inadequate family or caregiver support as determined by the site PI.
9. Presence of any of the following conditions:

   1. Current drug abuse or alcoholism
   2. Unstable medical conditions
   3. Unstable psychiatric illness including psychosis and untreated major depression within 90 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Safety of use of [11C]CPPC in patients with ALS as assessed by adverse events | Up to 180 days after scan
  Safety of use of [11C]CPPC in positron emission tomography (PET) neuroimaging of patients with a diagnosis of ALS. Safety will be assessed by number of adverse events during and up to 180 days after the injection
Safety of use of [11C]CPPC in patients with ALS as assessed by a change in neurological status | Baseline and 180 days after scan
  Safety of use of [11C]CPPC in positron emission tomography (PET) neuroimaging of patients with a diagnosis of ALS. Safety will be assessed by neurological physical exam to determine if there is a change in the findings from baseline.
Safety of use of [11C]CPPC in patients with ALS as assessed by a change in complete blood count (CBC) test | Baseline and 180 days after scan
  Safety of use of [11C]CPPC in positron emission tomography (PET) neuroimaging of patients with a diagnosis of ALS. Safety will be assessed by monitoring of the complete blood count (CBC) for a change from baseline that is outside of the normal range.
Safety of use of [11C]CPPC in patients with ALS as assessed by a change in complete metabolic panel (CMP) test | Baseline and 180 days after scan
  Safety of use of [11C]CPPC in positron emission tomography (PET) neuroimaging of patients with a diagnosis of ALS. Safety will be assessed by a change in the CMP from baseline that is outside of the normal range.

SECONDARY OUTCOMES:
Sensitivity of use of [11C]CPPC as assessed by a radiologist | Up to 180 days after scan
  Sensitivity of use of [11C]CPPC in PET neuroimaging to detect ALS will be determined by comparing the PET images from patients with ALS with those from healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Maragakis, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No